CLINICAL TRIAL: NCT00406185
Title: Database Registry of the Intermountain Heart Collaborative Study
Status: Active, not recruiting | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 128-db1
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Coronary Artery Disease; Electrophysiology; Cardiovascular Disease
Keywords: Registry; cardiac catheterization laboratory; coronary heart disease; cardiovascular disease
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the registry is to collect and analyze clinical and laboratory data and tissue samples from patients who are diagnosed with any type of heart disease and to collect the same information and samples from healthy controls in participating Intermountain Healthcare facilities.

DETAILED DESCRIPTION:
This is a registry (database) project; there are no investigational treatments, drug or procedures associated with participation in registry activities. This project is an organized data gathering and storing (database) endeavor with specific focus on the precursors, modifiers, biological, and genetic parameters of heart disease and related medical conditions. Data collection will not immediately influence the course of treatment for any patient.Sample testing and data utilization for basic science, clinical, and epidemiologic and publication projects can be initiated using the databank.

The registry will enable researchers to determine best medical practices for predicting, preventing, and treating heart disease. The registry will: 1) develop standard methods to collect data and specimens which will be used for research to characterize patients diagnosed with heart disease as well as healthy controls and to assess differences in demographics and patient outcomes in both populations; 2) collect, process, and store patients' clinical data and tissue/blood samples; 3) analyze data collected; 4) use these resources to identify genes, genetic polymorphisms, genetic mutations, clinical methods and procedures, and/or biomarkers that predict, prevent, or treat heart disease and/or are associated correlate with lifestyle or disease outcomes; 5) publish and disseminate results.

ELIGIBILITY:
Inclusion Criteria:

1. The patient (male or non-pregnant female) must be > 18 years of age.
2. The patient or legally authorized representative must sign a written informed consent, prior to the procedure, using a form that is approved by the local Institutional Review Board.

Exclusion Criteria:

1. Neither patient nor patient representative understands spoken English.
2. Neither patient nor the patient's personal representative is willing to give written consent for participation.
3. Healthy control patients must sign their own consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing a procedure within the catheterization laboratory
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 1994-10; Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Outcome Risk | 30 years
  To evaluate risk factors, characteristics, and treatments to cardiovascular outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Joseph B Muhlestein, MD, Principal Investigator — Intermountain Healthcare, LDS Hospital
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

REFERENCES:
- [Background] Taylor GS, Muhlestein JB, Wagner GS, Bair TL, Li P, Anderson JL. Implementation of a computerized cardiovascular information system in a private hospital setting. Am Heart J. 1998 Nov;136(5):792-803. doi: 10.1016/s0002-8703(98)70123-1. PMID 9812073
- [Derived] Lappe JM, Horne BD, Shah SH, May HT, Muhlestein JB, Lappe DL, Kfoury AG, Carlquist JF, Budge D, Alharethi R, Bair TL, Kraus WE, Anderson JL. Red cell distribution width, C-reactive protein, the complete blood count, and mortality in patients with coronary disease and a normal comparison population. Clin Chim Acta. 2011 Nov 20;412(23-24):2094-9. doi: 10.1016/j.cca.2011.07.018. Epub 2011 Jul 27. PMID 21821014
- [Derived] Horne BD, May HT, Kfoury AG, Renlund DG, Muhlestein JB, Lappe DL, Rasmusson KD, Bunch TJ, Carlquist JF, Bair TL, Jensen KR, Ronnow BS, Anderson JL. The Intermountain Risk Score (including the red cell distribution width) predicts heart failure and other morbidity endpoints. Eur J Heart Fail. 2010 Nov;12(11):1203-13. doi: 10.1093/eurjhf/hfq115. Epub 2010 Aug 12. PMID 20705688
- [Derived] Horne BD, May HT, Muhlestein JB, Ronnow BS, Lappe DL, Renlund DG, Kfoury AG, Carlquist JF, Fisher PW, Pearson RR, Bair TL, Anderson JL. Exceptional mortality prediction by risk scores from common laboratory tests. Am J Med. 2009 Jun;122(6):550-8. doi: 10.1016/j.amjmed.2008.10.043. PMID 19486718
- [Derived] Horne BD, May HT, Anderson JL, Kfoury AG, Bailey BM, McClure BS, Renlund DG, Lappe DL, Carlquist JF, Fisher PW, Pearson RR, Bair TL, Adams TD, Muhlestein JB; Intermountain Heart Collaborative Study. Usefulness of routine periodic fasting to lower risk of coronary artery disease in patients undergoing coronary angiography. Am J Cardiol. 2008 Oct 1;102(7):814-819. doi: 10.1016/j.amjcard.2008.05.021. Epub 2008 Jul 10. PMID 18805103
- [Derived] Horne BD, Camp NJ, Anderson JL, Mower CP, Clarke JL, Kolek MJ, Carlquist JF; Intermountain Heart Collaborative Study Group. Multiple less common genetic variants explain the association of the cholesteryl ester transfer protein gene with coronary artery disease. J Am Coll Cardiol. 2007 May 22;49(20):2053-60. doi: 10.1016/j.jacc.2007.02.039. Epub 2007 May 4. PMID 17512363